CLINICAL TRIAL: NCT04470141
Title: A Phase II, Multicenter Study to Investigate the Efficacy and Safety of SHC014748M in Patients With Relapsed or Refractory Peripheral T Cell Lymphoma
Brief Title: A Study of SHC014748M in Patients With Relapsed or Refractory Peripheral T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHC014-II-02
Record Dates: First submitted 2020-06-29; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: PTCL; SHC014748M; Phosphatidylinositol 3-kinase (PI3K)
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHC014748M treatment (Experimental): SHC014748M capsule, 200mg QD, 28 days for each cycle
  Interventions: Drug: SHC014748M treatment

INTERVENTIONS:
Drug: SHC014748M treatment — Each treatment cycle is comprised of 28-day consecutive dosing of SHC014748M, 200mg QD (Days 1 to28). Upon completion of each cycle, patients may continue to receive oral SHC014748M if they can benefit from the treatment and the toxicity is tolerable.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SHC014748M in patients with relapsed or refractory relapsed or refractory Peripheral T Cell Lymphoma.

DETAILED DESCRIPTION:
This is a phase II, multicenter study to assess the efficacy and safety of SHC014748M, an oral inhibitor of PI3K delta, in patients with relapsed or refractory peripheral T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Adult, male and female volunteers, above 18 years of age inclusive.
* Histologically or cytologically confirmed diagnosis of relapsed or refractory Peripheral T Cell Lymphoma,including but not limited to peripheral T-cell lymphoma-unspecified(PTCL-U),angioimmunoblastic T-cell lymphoma(AITL),ALK+/ALK-anaplastic large cell lymphoma(ALCL),subcutaneous panniculitis-like T-cell lymphoma(SPTL). Eligible patients have failed or progressed at least one standard treatment, have no standard treatment, or are intolerant for standard treatment at this stage as determined by the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
* Life expectancy ≥ 3 months.
* Patients have at least 1 measurable lesion that measures ≥1.5 cm in a single dimension as assessed by CT or MRI.
* Adequate organ function, as defined by the following values:ANC≥1.0×10^9/L;PLT≥50×10^9/L;Hb≥80 g/L;TBIL≤2×ULN(TBIL>2×ULN for subjects with Gilbert syndrome,TBIL>3×ULN for subjects with focal compression of bile duct as determined by investigators);ALT and AST≤2.5×ULN(ALT and AST≤5×ULN for subjects with impaired liver function caused by hepatic infiltration as determined by investigators);CLcr> 50 mL/min(according to Cockcroft-Gault).
* Men and women of childbearing potential are willing to employ an effective method of contraception for the entire duration of study and 6 months after the last dose, and female subjects of childbearing potential have a negative pregnancy test at baseline.
* Volunteers did not participate in other clinical trials within 1 month prior to study entry.
* Provision of signed and dated, written informed consent prior to any study-specific evaluation.

Exclusion Criteria:

* Previous treatment with any PI3Kδ inhibitors.
* Had any other anti-tumor treatment within 4 weeks prior to screening(including radiotherapy, chemotherapy, Chinese herbal anti-tumor treatment and major surgery); targeted therapy with 5 half-life period prior to the first dose of study drug.
* Evidence of central nervous system involvement of the malignancy,including invasion of brain parenchyma and meninges, or spinal cord compression.
* Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, uncontrolled pleural effusion and ascites, uncontrolled diabetes, severe or debilitating lung disease.
* Have moderate or severe cardiac disease, including but not limited to severe arrhythmias or abnormal cardiac conduction, such as ventricular arrhythmias requiring clinical intervention, degree II-III atrioventricular block,QTcF≥450 ms for male, QTcF≥470 ms for female, or other structural heart disease with high risk as determined by investigators;history of acute coronary syndrome, congestive heart failure,aortic dissection,stroke or other≥grade 3 cardiovascular and cerebrovascular events within 6 months prior to the first dose of study drug;New York Heart Association (NYHA) Class II or greater heart failure, or LVEF<55%;uncontrolled hypertension(systolic blood pressure>180 mmHg or diastolic blood pressure>100 mmHg with two measurements in a row);any risk factors to increase QTc or arrhythmias, including heart failure,hypokalemia,congenital long QTc syndrome,family history of long QT interval syndrome or history of unexplained sudden death occurred in first degree relative less than 40 years of age, or using any concomitant medication known to produce QTc prolongation.
* Evidence of active bacterial, fungal, or viral infection, and need systemic treatment with one week prior to the first dose of study drug.
* Infection with hepatitis B virus(HBV) ( volunteers with HBsAg positive but HBV-DNA negative, or volunteers with HCV antibody positive but HCV-RNA negative can be enrolled), hepatitis C virus(HCV), syphilis,or human immunodeficiency virus (HIV).
* Have systematic hormonal therapy(prednisone>20mg/d or similar drugs with equivalent dose)or immunosuppressor therapy with 14 days prior to the first dose of study drug, except using topical,ocular,intra-articular,intranasal,inhaled corticosteroids,and preventive therapy using corticosteroids in short period(for instance,to prevent hypersensitivity to contrast media).
* Concomitant use of any strong inhibitors or inducers of CYP3A4(except drug withdrawal prior to the first dose of study drug).
* History of immune deficiency(acquired and congenital), or history of organ transplantation, or allogeneic bone marrow or hematopoietic stem cell transplantation; with active autoimmune disease or history of autoimmune disease including Interstitial pneumonia, autoimmune enteritis, autoimmune hepatitis and systemic lupus erythematosus.
* Prior autologous hematopoietic stem cell transplantation within 2 months prior to the first dose of study drug.
* History of any uncured malignant tumor in the past five years except for the following: clinically cured cervical or breast carcinoma in situ, local basal cell or squamous cell carcinoma of the skin, thyroid tumor.
* Severe gastrointestinal disease affecting ingesting, transporting and absorbing of the study drug, include inability to swallow the drug,malabsorption syndrome,uncontrollable nausea and vomiting,history of extensive gastrointestinal resection,uncurable recurrent diarrhea,atrophic gastritis(age of onset<60),uncurable severe gastric diseases,crohn's disease,ulcerative colitis or complete Intestinal obstruction.
* Adverse events occurred during previous anticancer therapy have not been recovered to ≤1(CTCAE 5.0)except toxicity with no significant risk determined by investigators such as alopecia.
* History of hypersensitivity to the main composition or any inactive excipient of the study drug.
* Women who are breastfeeding.
* With basic medical condition leading to risk of taking study drugs judged by investigators, or with confusion to toxicity and adverse events.
* Judgment by the investigator that the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 12 months

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | up to 12 months
Progression-Free Survival(PFS) | up to 12 months
Time to Response(TTR) | up to 12 months
Duration of Response(DOR) | up to 12 months
Mean Change From Baseline in the Functional Assessment of Cancer Therapy Lymphoma (FACT-Lym) Scale. | up to 12 months
  The FACT-Lym questionnaire is a validated instrument for assessing the impact of lymphoma on health related quality of life(HRQL) and contains 42 questions covering HRQL and common lymphoma symptoms and treatment side-effects. It begins with the Functional Assessment of Cancer Therapy - General (FACT-G), which contains 27 questions covering four core subscales: Physical Wellbeing (7 items), Social/Family Wellbeing (7), Emotional Wellbeing (6), and Functional Wellbeing (7). The FACT-Lym also includes an Additional Concerns subscale (15 questions) used to assess non-Hodgkins lymphoma(NHL) related symptoms and concerns. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). Higher scores are associated with a better quality of life.
Safety and Tolerability of SHC014748M Assessed as the Number of Participants Experiencing Adverse Events (AEs) or Abnormalities in Vital Signs, Laboratory Tests, or Electrocardiograms. | up to 12 months